CLINICAL TRIAL: NCT01772693
Title: A Feasibility Study to Evaluate Safety and Initial Effectiveness of ExAblate Transcranial MR Guided Focused Ultrasound for Unilateral Thalamotomy in the Treatment of Medication-Refractory Tremor Dominant Idiopathic Parkinson's Disease.
Brief Title: ExAblate Transcranial MR Guided Focused Ultrasound for the Treatment of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PD001
Record Dates: First submitted 2012-11-28; First posted 2013-01-21 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-07

CONDITIONS: Parkinson's Disease
Keywords: ExAblate Transcranial MRgFUS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Single factor. ExAblate test verses ExAblate placebo randomized 2:1.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ExAblate Transcranial MRgFUS (Experimental): ExAblate Transcranial MR guided Focused Ultrasound
  Interventions: Device: ExAblate Transcranial MRgFUS
- Sham ExAblate Transcranial MRgFUS (Sham Comparator): Sham treatment with ExAblate MR guided Focused Ultrasound
  Interventions: Device: Sham ExAblate Transcranial MRgFUS

INTERVENTIONS:
Device: ExAblate Transcranial MRgFUS — ExAblate Transcranial MR Guided Focused Ultrasound
  Other Names: ExAblate; MRgFUS; Focused Ultrasound; Transcranial MRgFUS Thalamotomy
  Arms: ExAblate Transcranial MRgFUS
Device: Sham ExAblate Transcranial MRgFUS — Sham ExAblate Transcranial MR Guided Focused Ultrasound
  Arms: Sham ExAblate Transcranial MRgFUS

SUMMARY:
This is a feasibility study to evaluate the safety and initial effectiveness of unilateral ExAblate thermal ablation of the Vim thalamic nucleus of subjects suffering from medication-refractory, idiopathic, tremor-dominant PD, using the ExAblate Transcranial system compared to a Sham Vim thalamotomy procedure.

Data will be collected to establish the basic safety of this type of treatment as the basis for later studies that will evaluate its full clinical efficacy. The Sham treatment data will be used to evaluate placebo effect from treatment.

DETAILED DESCRIPTION:
Subjects who sign informed consent and pass all eligibility criteria will be randomized to a treatment assignment. During treatment, the assigned treatment (ExAblate Transcranial or Sham ExAblate Transcranial)will be delivered. Subjects are followed in a blinded fashion for three (3) months. After the 3-month assessment, subjects will be unblinded and told their treatment assignment. Subjects receiving Sham ExAblate Transcranial treatment who still meet criteria will be crossed over and receive an active ExAblate Transcranial treatment. Subjects will be followed for up to two (2) years. Follow-up at 1 week, 1 month, 3 months, 6 months, 9 months, 12 months and up to two (2) years includes Unified Parkinson's Disease Rating Scale (UPDRS) scoring, mental and cognitive functional testing and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 30 years and older
* Subjects who are able and willing to give informed consent and able to attend all study visits
* Subjects with a diagnosis of idiopathic PD as confirmed from clinical history and examination by a movement disorder neurologist at the site
* Subject demonstrates a severe resting tremor or postural/action as measured by UPDRS
* Subject exhibits a significant disability from their PD tremor despite medical treatment
* Subjects should be on a stable dose of all PD medications for 30 days prior to study entry
* Subject is able to communicate sensations during the ExAblate Transcranial procedure

Exclusion Criteria:

* Subjects with unstable cardiac status
* Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse
* Severe hypertension
* Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
* Known intolerance or allergies to the MRI contrast agent including advanced kidney disease or severely impaired renal function
* Significant claustrophobia that cannot be managed with mild medication
* Current medical condition resulting in abnormal bleeding and/or coagulopathy
* Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage
* History of intracranial hemorrhage
* History of multiple strokes, or a stroke within past 6 months
* Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment
* Are participating or have participated in another clinical trial in the last 30 days
* Subjects unable to communicate with the investigator and staff
* Subjects with a history of seizures within the past year
* Subjects with brain tumors
* Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment
* Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Elias, M.D., Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - University of Virginia, Charlottesville, Virginia
  - Swedish Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Bond AE, Shah BB, Huss DS, Dallapiazza RF, Warren A, Harrison MB, Sperling SA, Wang XQ, Gwinn R, Witt J, Ro S, Elias WJ. Safety and Efficacy of Focused Ultrasound Thalamotomy for Patients With Medication-Refractory, Tremor-Dominant Parkinson Disease: A Randomized Clinical Trial. JAMA Neurol. 2017 Dec 1;74(12):1412-1418. doi: 10.1001/jamaneurol.2017.3098. PMID 29084313

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ExAblate Transcranial MRgFUS | Sham ExAblate Transcranial MRgFUS
Started | 20 | 7
Completed | 14 | 6
Not Completed | 6 | 1
Not completed — Health Concerns Unrelated to Study | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Alternative Treatment | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ExAblate Transcranial MRgFUS | Sham ExAblate Transcranial MRgFUS | Total
Number analyzed (Participants) | 20 | 7 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (9.6) | 62.9 (11.3) | 66.6 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 19 | 7 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 18 | 6 | 24
  Race: Black | 2 | 0 | 2
  Race: Other | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 7 | 27
Clinical Rating Scale for Tremor - Treated Side [Mean (Standard Deviation); unit: units on a scale] — Baseline sum of upper extremity Tremor-Motor scores for the treated side from the Clinical Rating Scale for Tremor (CRST) Part A and Part B averaged across subjects. This measure of upper extremity tremor ranges from 0-32 with high scores being worse.
  units on a scale | 19.0 (8.7) | 20.1 (7.4) | 19.3 (8.3)
Mean Unified Parkinson's Disease Rating Scale (UPDRS) #20 [Mean (Standard Deviation); unit: units on a scale] — The Unified Parkinson's Disease Rating Scale (UPDRS) Question 20 is a measure of tremor of the treated side hand at rest on a score from 0 to 4 points. High scores are worse. Scores are averaged across subjects.
  units on a scale | 3.7 (1.0) | 3.4 (1.5) | 3.6 (1.1)
Mean Unified Parkinson's Disease Rating Scale (UPDRS) #21 [Mean (Standard Deviation); unit: units on a scale] — The Unified Parkinson's Disease Rating Scale (UPDRS) Question 21 is an assessment of action or postural tremor of the treated side hand scored from 0 to 4. High scores are worse. The scores are averaged across subjects.
  units on a scale | 3.2 (1.3) | 3.6 (1.1) | 3.3 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Description: Evaluate of adverse events (AEs) associated with the ExAblate Transcranial thalamotomy of medication-refractory, tremor-dominant PD during the ExAblate treatment.
  Primary safety analyses are reported in the adverse events module.
Time Frame: Month 3
Population: All Adverse Events are reported in the Adverse Events module.
Measure: Number; unit: Number of Adverse Events
Arm/Group | ExAblate Transcranial MRgFUS | Sham ExAblate Transcranial MRgFUS
Number analyzed (Participants) | 20 | 7
Number of Adverse Events | 100 | 10

2. Secondary Outcome: Tremor Motor Score Percent Change From Baseline.
Description: The percent change from baseline to Month 3 follow-up in upper extremity Tremor-Motor scores for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum that was used to measure treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points. Individual subject's scores at Baseline and 3 Months were used to calculate percent change from baseline and averaged across subjects. High percent change from baseline is better (shows improvement).
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: percent change from baseline
Arm/Group | ExAblate Transcranial MRgFUS | Sham ExAblate Transcranial MRgFUS
Number analyzed (Participants) | 20 | 7
percent change from baseline | 51.9 (33.4) | 12.7 (25.7)

3. Secondary Outcome: Tremor Motor Scores - Clinical Rating Scale for Tremor - Treated Side Upper Extremity Parts A & B.
Description: Upper extremity Tremor-Motor score for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum that measures treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points for each side with lower scores being a better outcome. Subject's Tremor-Motor scores for the test and sham control groups were averaged at each study visit.
Time Frame: Baseline, Month 3, Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ExAblate Transcranial MRgFUS | Sham ExAblate Transcranial MRgFUS
Number analyzed (Participants) | 20 | 7
score on a scale
  Baseline | 19.0 (8.7) | 20.1 (7.4)
  Month 3 | 9.6 (9.7) | 17.4 (7.8)
  Month 12 | 10.5 (10.2) | NA (NA) — The sham ExAblate subjects exited the study at Month 3. The Exablate test subjects continued through Month 12.

4. Secondary Outcome: Functional Disabilities - Clinical Rating Scale for Tremor Part C - Functional Disabilities
Description: The Clinical Rating Scale for Tremor (CRST) Part C is a measure of functional disability due to tremor. The Clinical Rating Scale for Tremor Part C consists of 8 items each scored from 0 to 4. Thus, the total score summed ranges from 0 to 32 and provides an overall assessment of activities of daily living. Low scores on the Clinical Rating Scale for Tremor (CRST) Part C are better. Low scores show improvement in functional disabilities compared to higher scores.
Time Frame: Baseline, Month 3, Month 12
Population: The Exablate sham subjects exited the study at the Month 3 visit. The Exablate test subjects continued on through Month 12.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ExAblate Transcranial MRgFUS | Sham ExAblate Transcranial MRgFUS
Number analyzed (Participants) | 20 | 7
score on a scale
  Baseline | 14.1 (5.7) | 16.7 (3.9)
  Month 3 | 6.4 (6.6) | 14.6 (4.2)
  Month 12 | 6.9 (7.2) | NA (NA) — The Exablate sham subjects exited the study at the Month 3 study visit.

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | ExAblate Transcranial MRgFUS | Sham ExAblate Transcranial MRgFUS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/20 | 1/7
Other Adverse Events (participants affected / at risk) | 20/20 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Transcranial MRgFUS (N=20) | Sham ExAblate Transcranial MRgFUS (N=7)
Hemiparesis (Nervous system disorders) | 2 (2) | 0 (0) — After Focused Ultrasound Surgery thalamotomy procedure. Determined event to be SAE related to thalamotomy.
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) — Event 1 component was mild right-sided hemiparesis (weakness) with drift. Event expected and related to thalamotomy. Resolved.
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated to device or procedure
Degenerative knee disease (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated to device or procedure. Subject had knee replacement and physical therapy. Adverse event resolved.
Worsening depression (Psychiatric disorders) | 1 (1) | 0 (0) — Since his tremor was gone he stopped his dopamine antagonist and he also stopped his antidepressants. His physicians planned to re-instate antidepressant medications and neuropsychology treatment.
Transient ischemic attack (Vascular disorders) | 0 (0) | 1 (1) — The Data Safety Monitoring Board discussed the event, the subject's symptoms and the lack of imaging findings and determined that they agreed with the investigator that this event was Unrelated to the Exablate procedure.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Transcranial MRgFUS (N=20) | Sham ExAblate Transcranial MRgFUS (N=7)
Sleep Disorder (General disorders) | 1 (1) | 0 (0) — Related to Parkinson's Disease progression.
Dysgnosia (Nervous system disorders) | 0 (0) | 1 (1) — Related to Parkinson's Disease progression
Tremor worsened (Nervous system disorders) | 1 (1) | 0 (0) — Related to Parkinson's Disease progression
Fatique (General disorders) | 2 (2) | 0 (0) — Procedure related
Musculoskeletal weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Procedure related
Dysgnosia (Nervous system disorders) | 1 (1) | 0 (0) — Procedure related
Dizziness (Ear and labyrinth disorders) | 1 (1) | 1 (1) — Procedure related
Dysmetria (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Thalamotomy related
Gait disturbance (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) — Thalamotomy related
Hemiparesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Imbalance (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) — Thalamotomy related
Dysmetria (Nervous system disorders) | 2 (2) | 0 (0) — Thalamotomy related
Ataxia (Nervous system disorders) | 2 (2) | 0 (0) — Thalamotomy related
Numbness/tingling (Nervous system disorders) | 7 (8) | 0 (0) — Thalamotomy related
Unsteady (Nervous system disorders) | 1 (1) | 0 (0) — Thalamotomy related
Hypertension (Vascular disorders) | 1 (1) | 0 (0) — Transient
Syncope (Vascular disorders) | 1 (1) | 0 (0) — Transient
Sonication related flushing (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Transient
Visual field defect (Eye disorders) | 1 (1) | 0 (0) — Transient
Nausea/Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1) — Transient
Imbalance (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Transient
Positional pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) — Transient
Imbalance (Nervous system disorders) | 1 (1) | 0 (0) — Transient
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) — Transient
Dysgnosia (Psychiatric disorders) | 2 (2) | 0 (0) — Transient
Numbness/tingling (Nervous system disorders) | 5 (7) | 0 (0) — Transient
Headache (General disorders) | 11 (11) | 2 (2) — Transient
Sonication related scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Transient
Sonication related head pain (General disorders) | 5 (6) | 1 (1) — Transient
Pin Site Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Transient
Dizziness (Ear and labyrinth disorders) | 7 (7) | 0 (0) — Transient
Pigment change in eye (Eye disorders) | 1 (1) | 0 (0) — Unrelated
Vision change (Eye disorders) | 1 (1) | 0 (0) — Unrelated
Cholecystitis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Unrelated
Vocal change (General disorders) | 1 (1) | 0 (0) — Unrelated
Worsening depression (Psychiatric disorders) | 1 (1) | 0 (0) — Unrelated
Musculoskeletal weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) — Unrelated
Positional pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Unrelated
Cerebelar infarct (Vascular disorders) | 1 (1) | 0 (0) — Unrelated
Dizziness (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Unrelated
Transient Ischemic Attack (Vascular disorders) | 0 (0) | 1 (1) — Unrelated
Facial edema (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) — Unrelated
Pin site numbness/tingling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Unrelated
Pin site pain (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) — Unrelated
Stereotactic frame bruising (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Unrelated

LIMITATIONS AND CAVEATS:
This is a feasibility trial with no pre-defined hypothesis testing. It is primarily a safety trial with a secondary objective of collecting efficacy outcomes for developing future pivotal trials.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No